CLINICAL TRIAL: NCT00852852
Title: Computerized Assessment for Patients With Cancer-ESRA-C II
Brief Title: Computerized Assessment for Patients With Cancer
Acronym: ESRA-C_II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); University of Washington (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Donna Berry, PhD, RN, FAAN, AOCN, Assoc. Professor, Harvard Medical School; Director, The Phyllis F. Cantor Center, Research in Nursing and Patient Care Services; Affiliate Professor, University of Washington School of Nursing, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-284; R01NR008726 (NIH)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Cancer
Keywords: ESRA-C 2; computerized assessment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Patient participants in the intervention arm can access educational information about self-care strategies, track and share reports of their symptoms and quality of life issues over time, and receive coaching on how to discuss these issues with their care team.
  Interventions: Behavioral: Electronic Self-Report Assessment - Cancer (ESRA-C)
- Control (No Intervention): Participants in the control arm access the ESRA-C from home or clinic to self-assess only.

INTERVENTIONS:
Behavioral: Electronic Self-Report Assessment - Cancer (ESRA-C) — The Electronic Self-Report Assessment-Cancer (ESRA-C) is a program allowing patients to report symptoms and quality of life issues and learn information about how to deal with these experiences.
  Arms: Intervention

SUMMARY:
This research study will test a new online computer program for patients, the Electronic Self-Report Assessment-Cancer (ESRA-C 2). The program allows patients to report symptoms and quality of life issues and learn information about how to deal with these experiences. The computer program is being tested to see if it can improve communications between patients and their care team and if it can improve patients' experiences during and after treatment.

DETAILED DESCRIPTION:
* This study includes two groups of participants: 1) Clinician Participants and 2) Patient Participants.
* Patient participants will have already completed one ESRA-C 2 report, which is a usual report in the clinic. If they decide to participate in the study, that report will be used in the study as the first report (Timepoint 1). In addition, they will complete a second report (Timepoint 2) and two more reports (Timepoint 3 and 4). Timepoint 3 will be 6-8 weeks after the participants treatment begins; Timepoint 4 will be 2-4 weeks after their treatment ends.
* The Timepoint 2 report will be within 24 hours before a clinic visit. The conversation between the patient participant and the health care providers will be audio recorded.
* Half of the patient participants will also see additional information in the computer program. The patient participants that are in this group can complete as many more ESRA-C 2 reports as they wish and will be able to read additional information about managing symptoms and quality of life issues, view graphs of their reports, add journal entries, and share all their reports with caregivers.
* Clinician Participants will be asked to report brief demographics (age group, gender, race/ethnicity, position). During clinic appointments, research staff will place a 3" by 5" audio-recorder in the exam room just prior to some of the participant's visits. Recordings will be de-identified before coding.
* After these visits, a research staff member will ask the clinician participant to report briefly on their satisfaction in the visit. The participant can check their responses on a piece of paper or dictate them.

ELIGIBILITY:
Eligible clinician participants (Inclusion):

* Nurses, physicians, or physician assistants
* Perform consults/exams in clinics that have implemented routine use of the ESRA-C 2 screening tool as a standard of care

Eligible patient participants (Inclusion):

* 18 years of age or older
* Diagnosis of malignant disease
* Plan to have treatment in a study clinic
* Speak and read English at a 6th grade level or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Symptom burden and quality of life 2-4 weeks post treatment | 3 years

SECONDARY OUTCOMES:
To assess the feasibility of delivering a patient oriented, patient-controlled ESRA-C directly to patients outside clinically settings. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Donna L. Berry, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knoerl R, Hong F, Blonquist T, Berry D. Impact of Electronic Self-Assessment and Self-Care Technology on Adherence to Clinician Recommendations and Self-Management Activity for Cancer Treatment-Related Symptoms: Secondary Analysis of a Randomized Controlled Trial. JMIR Cancer. 2019 Jan 8;5(1):e11395. doi: 10.2196/11395. PMID 30622093
- [Derived] Knoerl R, Weller E, Halpenny B, Berry D. Exploring the efficacy of an electronic symptom assessment and self-care intervention to preserve physical function in individuals receiving neurotoxic chemotherapy. BMC Cancer. 2018 Dec 4;18(1):1203. doi: 10.1186/s12885-018-5093-z. PMID 30514351
- [Derived] Siefert ML, Bonquist TM, Berry DL, Hong F. Symptom-related emergency department visits and hospital admissions during ambulatory cancer treatment. J Community Support Oncol. 2015 May;13(5):188-94. doi: 10.12788/jcso.0134. PMID 27119127
- [Derived] Berry DL, Blonquist TM, Patel RA, Halpenny B, McReynolds J. Exposure to a patient-centered, Web-based intervention for managing cancer symptom and quality of life issues: impact on symptom distress. J Med Internet Res. 2015 Jun 3;17(6):e136. doi: 10.2196/jmir.4190. PMID 26041682
- [Derived] Berry DL, Hong F, Halpenny B, Partridge A, Fox E, Fann JR, Wolpin S, Lober WB, Bush N, Parvathaneni U, Amtmann D, Ford R. The electronic self report assessment and intervention for cancer: promoting patient verbal reporting of symptom and quality of life issues in a randomized controlled trial. BMC Cancer. 2014 Jul 12;14:513. doi: 10.1186/1471-2407-14-513. PMID 25014995
- [Derived] Hong F, Bosco JL, Bush N, Berry DL. Patient self-appraisal of change and minimal clinically important difference on the European organization for the research and treatment of cancer quality of life questionnaire core 30 before and during cancer therapy. BMC Cancer. 2013 Mar 28;13:165. doi: 10.1186/1471-2407-13-165. PMID 23537330